## Statistical analysis

All statistical analyses were performed using SPSS for Windows version 21.0 (IBM SPSS, Armonk, NY: IBM Corp.). Continuous variables were given as mean  $\pm$  standard deviation, and categorical variables as numbers (n) and percent (%). The relationship between QoL and other parameters was tested with Spearman Correlation Analysis because not normally distributed continuous variables, after testing variables for normality using the Shapiro-Wilk test. Mann-Whitney U test was used to compare PD patients who with and without tremor. Significance level was accepted as p<0.05.